CLINICAL TRIAL: NCT02661841
Title: Effectiveness of Lung Impedance Guided Preemptive Therapy of Chronic Heart Failure Patients With Preserved Ejection Fraction (LVEF ≥ 45%) in Our Hospital's Outpatient Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0086-15 HYMC
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LI-Guided Therapy (Experimental): One hundred and fifty chronic heart failure patients treated based on guidelines and LI-Guided Therapy.
  Interventions: Other: LI-Guided Therapy; Other: Heart Failure Guidelines
- Control (Active Comparator): One hundred and fifty chronic heart failure patients treated based on guidelines only.
  Interventions: Other: Heart Failure Guidelines

INTERVENTIONS:
Other: LI-Guided Therapy — Preemptive treatment according to LI monitoring
  Arms: LI-Guided Therapy
Other: Heart Failure Guidelines — Treatment according to clinical signs

SUMMARY:
We aim to determine the effectiveness of lung impedance guided preemptive therapy (LI-Guided) of chronic heart failure patients with preserved ejection fraction (LVEF ≥ 45%) who are being treated in our hospital's outpatient clinic.

DETAILED DESCRIPTION:
Protocol Impedance HFpEF study Eligible patients are: older than 18 years, had a left ventricle ejection fraction (LVEF) > 45% with New York Heart Association (NYHA) functional class II-IV, and have been hospitalized for Heart Failure within 12 months of recruitment . The study requires optimal medical therapy for HF according to current guidelines. Patients have to be followed for at least 12 months. Exclusion criteria are: implantation of a cardiac resynchronization device within the preceding 3 months and the presence of advanced chronic kidney disease (estimated glomerular filtration rate <25 mL/min per 1.73 m2). All patients provided written informed consent. Randomization is: 1:1 to the active LI-guided treatment arm where clinicians are unblinded to LI values and could base therapy on LI level during outpatient clinic visits. In the control arm LI values are recording but not conveying to the clinical treatment team. In the case of hospitalization, LI is also recorded but this information was not provided to the treating physician. However, once patients resumed in hospital care LI was again provided to the treatment team only if the patient is assigned to the actively LI-guided group.

Inpatient study protocol At each out hospital visit such parameters as: vital signs, weight, jugular venous pressure (JVP), leg edema (0-4 points according to the level of lower limb edema), extent of lung rales (0- no rales, 1- basilar rales, 2- up to 1/3 of the lower lung field, 3- up to 1/2 of the lower lung field, 4- rales beyond half of the lung field) and oximetry were recorded, and NYHA class assessed. Chest radiographs (CXR) were performed at hospital admission and discharge. JVP was graded according to a modified Evaluation Study of Congestive Heart Failure and Pulmonary Artery Catheterization Effectiveness (ESCAPE) trial scale, i.e., maximal level of venous pulsation above sternal angle < 3 cm was defined as JVP= 0, a level of 3-5 cm as JVP= 1, 5-8 cm as JVP= 2, 8-11 cm as JVP = 3 and level of venous head> 11 cm as JVP = 4 are registered. NT-pro BNP level is measured at admission and discharge. CXRs and NT-pro BNP samples were used to substantiate the cause of admission, the degree of pulmonary congestion and extent of improvement during hospitalization. The 10-point radiological score (RS) was applied to assess the CXR when RS=0 signifies no congestion; RS of 1-4 represents interstitial congestion; and RS of 5-10 is compatible with alveolar edema. Medical therapy administered during hospitalization has to be documented.

This information is correct up to December 31, 2017. To date, there have been 24 participants in the interventional arm of the study and 24 in the control group.

Study update June 17, 2020: To date we have enrolled 102 patients (51 patients in each arm). The data monitoring committee of the study has reviewed the ongoing results and has allowed its continuation to the following year.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized within past 12 months for heart failure

Exclusion Criteria:

* Dialysis patients
* Patients with GFR <25
* Patients with serious illness and life expectancy <12
* Mentally incompetent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Reduced all cause, cardiovascular, and heart failure hospitalizations | Five years
Reduced mortality | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shochat, MD, PhD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No